CLINICAL TRIAL: NCT01894529
Title: Clinical Implications of a Panel of Immunological Biomarkers in Patients With Acute Ischemic Stroke
Brief Title: Immunological Biomarkers in Patients With Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Angel Chamorro, M.D., Ph.D., Ángel Chamorro, Hospital Clinic of Barcelona
Other Study IDs: PI09/1313
Record Dates: First submitted 2013-07-04; First posted 2013-07-10 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; immune biomarkers; stroke-associated infection; functional outcome; prediction
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum and plasma.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ischemic stroke: Patients with an ischemic stroke admitted within 6 hours of symptom onset, with a minimum severity in the NIHSS of 3 and treated with systemic or intraarterial thrombolysis
- Healthy subjects: Age-matched individuals free of acute neurological injury

SUMMARY:
Stroke is accompanied by local inflammatory response and systemic immunosuppression. Immunosuppression markers are associated with the occurrence of medical complications (infections), whereas inflammatory markers are associated with worse functional prognosis.

This prospective study tries to validate in acute stroke patients the prognostic usefulness of a panel of immune biomarkers that have previously been associated with various clinical outcomes.

The identification of beneficial and harmful immune responses in cerebral ischemia will allow the prediction of the clinical course of the patients and will be helpful in designing immunomodulatory therapeutic strategies for acute stroke.

DETAILED DESCRIPTION:
Stroke is accompanied by local inflammatory response and systemic immunosuppression. Immunosuppression markers are associated with the occurrence of medical complications (infections), whereas inflammatory markers are associated with worse functional prognosis.

This prospective study tries to validate in acute stroke patients the prognostic usefulness of a panel of immune biomarkers that have previously been associated with various clinical outcomes. The immune biomarkers will be assessed at admission, at day 1 after admission and at day 90. The assessed immune biomarker panel includes:

* Serum cortisol levels.
* Serum interleukin (IL)-10 levels.
* Proportion of circulating B lymphocytes (CD3-CD19+ cells).
* Monocyte surface expression of TLR4, HLA-DR, CD86, and VLA-4.
* Ex - vivo production of tumor necrosis factor (TNF)-α in monocytes after stimulation with LPS.
* Proportion of each of the circulating monocyte subpopulations (CD14highCD16-, CD14highCD16+, and CD14dimCD16+).

The identification of beneficial and harmful immune responses in cerebral ischemia will allow the prediction of the clinical course of the patients and will be helpful in designing immunomodulatory therapeutic strategies for acute stroke.

ELIGIBILITY:
Inclusion Criteria:

* ischemic stroke*
* stroke onset within 6h*
* treated with systemic or intraarterial thrombolysis*
* minimum severity in the NIHSS of 3*
* age ≥ 18
* consent by the patient or the legal representative

  * These items do not apply for healthy subjects.

Exclusion Criteria:

* intracranial hemorrhage
* signs of infection at admission
* use of antibiotics, immunosuppressors or corticosteroids in the previous 3 months
* significant disability (mRS>2) before index stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with an ischemic stroke admitted within 6 hours of symptom onset, with a minimum severity in the NIHSS of 3 and treated with systemic or intraarterial thrombolysis and age-matched subjects free of acute neurological injury.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2010-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Predictive immune score for favorable outcome | 90 +-15 days after onset of symptoms
  To establish a predictive immune score for functional outcome. Favorable outcome is defined as a modified Rankin Scale (mRS) score of <3 at day 90+-15 after stroke
Predictive immune score for stroke associated infection | 7 days after onset of symptoms
  To establish a predictive score for stroke associated infection (SAI) based on immune biomarkers. Stroke associated infection is defined as: body temperature > 37.7ºC and symptoms of infection (cough, dyspnea, pleuritic pain, dysuria), or leukocytosis >11000, leukopenia <4000, pulmonary infiltrates in chest X-ray or positive cultures for a pathogen.

SECONDARY OUTCOMES:
Predictive immune score for ischemic progression | 7 days after onset of symptoms
  To establish a predictive score for ischemic progression based in a panel of immune biomarkers. Ischemic progression is defined as an increase of ≥4 points in the National Institutes of Health Stroke Scale(NIHSS) score in the absence of bleeding in the CT scan.
Predictive immune score for functional outcome over the entire mRS | 90 +-15 days after onset of symptoms
  To establish a predictive score for functional outcome based in a panel of immune biomarkers and using shift analysis of the entire mRS
Localization and stroke volume analysis | SAI within 7 days and neurological outcome after 3 months after onset of symptoms
  To investigate the influence of the localization and stroke volume on the occurrence of a stroke associated infection and on neurological outcome
Insular cortex involvement and infarct volume | SAI within 7 days and and on the neurological outcome after 3 months
  To investigate the influence of insular cortex involvement and infarct volume on the occurrence of a SAI and on the neurological outcome after 3 months
Infection and functional outcome after ischemic stroke | SAI within 7 days after onset of symptoms and neurological outcome after 3 months
  To assess the independent effect of SAI over the functional outcome at 3 months
Thrombolysis, immune biomarkers and SAI | SAI within 7 days after onset of symptoms
  To assess the effect of thrombolytic treatment over changes in the immune biomarker panel and over the occurrence of SAI

CONTACTS AND LOCATIONS:
Overall Officials: Angel Chamorro, MD, PhD, Principal Investigator — Functional Unit of Cerebrovascular Diseases (Hospital Clínic of Barcelona), IDIBAPS and University of Barcelona Barcelona, Spain
Locations (1):
- Functional Unit of Cerebrovascular Diseases, Hospital Clínic of Barcelona, Barcelona, Barcelona, Spain